CLINICAL TRIAL: NCT02258958
Title: Extended Out-of-hospital Low-molecular-weight Heparin Prophylaxis Against Deep Venous Thrombosis and Pulmonary Embolus in Patients Undergoing Major Lung Resection: A Pilot Study to Evaluate the Incidence of DVT and PE After Major Lung Resection
Brief Title: Extended Out-of-hospital Low-molecular-weight Heparin Prophylaxis Against DVT and PE in Patients Undergoing Major Lung Resection
Status: Completed | Type: Observational
Sponsor: McMaster University (Other)
Collaborators: Toronto General Hospital (Other); Heart and Stroke Foundation of Canada (Other)
Responsible Party: Principal Investigator, Yaron Shargall, Head of Services Thoracic Surgery, McMaster University
Other Study IDs: SJHH_VTEincidence; 13-368 (Other: Hamilton Integrated Research Ethics Board)
Record Dates: First submitted 2014-10-03; First posted 2014-10-08 (Estimated); Last update posted 2014-12-18 (Estimated); Status verified 2014-12

CONDITIONS: Venous Thrombosis; Pulmonary Embolism; Lung Neoplasms
Keywords: venous thromboembolism prophylaxis; deep venous thrombosis; pulmonary embolus; thoracic surgery; lung resection; incidence
MeSH Terms: conditions — Venous Thrombosis; Pulmonary Embolism; Lung Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Postoperative venous thromboembolism (VTE) is a significant health-care problem, resulting in significant morbidity, mortality and resource utilization. The true incidence is unknown, and may range from 1% to 15%. At the current time, the clinical practice of VTE prophylaxis in thoracic surgery includes administration of unfractionated or low molecular weight heparin starting at the perioperative period and finishing at the time of patients' discharge. In orthopaedic surgery, prolonged thromboprophylaxis beyond 10 days and up to 35 days has become the standard of care. There is a clear need to systematically evaluate the incidence of VTE after resection of lung malignancies and to evaluate the role of extended VTE prophylaxis in preventing Deep Vein Thrombosis (DVT) and pulmonary embolus (PE) after those major lung resections. This study will involve patients undergoing lung resection for malignancy at St. Joseph's Healthcare Hamilton and the University Health Network's Toronto General Hospital. The study will include 150 consecutively recruited patients. Study interventions will include Computed Tomography with pulmonary embolus (PE) protocol and bilateral extended leg Doppler Ultrasound for the detection of Deep Vein Thrombosis 30 days post-surgery.

In summary, this study is aimed at evaluating, for the first time in a prospective manner, the actual incidence of DVT and PE in patients undergoing major lung resections for malignancies. The knowledge gained in this study will be used to inform a future investigation involving a Randomized Controlled Trial (RCT) to compare current post-operative thromboprophylaxis with an extended 30-day prophylaxis protocol with the hope of providing an evidence-based practice change in VTE prophylaxis care for this high risk population.

DETAILED DESCRIPTION:
Postoperative venous thromboembolism (VTE) is a significant health-care problem, resulting in significant morbidity, mortality and resource utilization. The true incidence is unknown, and may range from 1% to 15%. The latest American College of Chest Physicians (ACCP) guidelines on VTE prevention clearly outlines the perioperative thromboprophylaxis regiments for specific surgical populations. Specifically for patients undergoing orthopaedic procedures, such as total hip replacement, there is strong Grade 1A evidence for the use of extended thromboprophylaxis. For other surgical subgroups such as vascular and thoracic surgery, the evidence is less clear.

Therefore at the current time, the clinical practice of VTE prophylaxis in thoracic surgery includes administration of unfractionated or low molecular weight heparin starting at the perioperative period and finishing at the time of patients' discharge. Prolonged thromboprophylaxis in orthopaedic surgery beyond 10 days and up to 35 days has become the standard of care and has Grade 1A recommendations from ACCP. This approach has never been tested or validated in thoracic surgery, where major lung resection exposes the patient to an increased VTE risk not only due to the surgical stress and existence of malignancy, but also due to direct in-situ vascular injury secondary to resection of pulmonary arterial branches during the lung resection. Hence, there is a clear need to systematically evaluate the incidence of VTE after resection of lung malignancies and to evaluate the role of extended VTE prophylaxis in preventing DVT and pulmonary embolus (PE) after those major lung resections.

The study will involve patients undergoing sub-lobar resection, lobectomy, bilobectomy or pneumonectomy for lung cancer or metastatic lung disease at St. Joseph's Healthcare Hamilton, a regional tertiary thoracic surgery program with more than 350 major lung resections performed within the institution annually, as well as the University Health Network's Toronto General Hospital. The study will evaluate the incidence of post-operative venous thromboembolism (VTE) and will include 150 consecutively recruited patients. Study interventions will include Computed Tomography with pulmonary embolus (PE) protocol and bilateral extended leg Doppler Ultrasound for the detection of Deep Vein Thrombosis 30 days post-surgery.

In summary, this study is aimed at evaluating, for the first time in a prospective manner, the actual incidence of DVT and PE in patients undergoing major lung resections for malignancies. The knowledge gained in this study will be used to inform a future investigation involving an RCT to compare current post-operative thromboprophylaxis with an extended 30-day prophylaxis protocol with the hope of providing an evidence-based practice change in VTE prophylaxis care for this high risk population.

ELIGIBILITY:
Patient Inclusion Criteria

* At least 18 years of age
* Either gender
* Diagnosed with resectable lung cancer or metastatic lung disease eligible to complete metastasectomy
* Undergoing one of the following surgeries: Segmentectomy, wedge resection, lobectomy, bilobectomy or pneumonectomy
* Competent to understand and sign consent documents

Patient Exclusion Criteria

* Known allergic or anaphylactic reaction to contrast dye, heparin or low molecular weight heparin (LMWH)
* Under current anticoagulation for venous thromboembolism or other medical conditions
* Known renal impairment, defined as creatinine clearance value of less than 55ml/min/m2 as calculated by the Cockroft-Gault method
* History of, or ongoing liver disease, manifested as ascites or previous peritoneal tapping for ascites
* Pregnant or planning to become pregnant
* Diagnosed or treated for VTE in the past 3 months prior to surgery
* Present or previous increase risk of haemorrhage
* History of previous HIT (heparin induced thrombocytopenia)
* Platelet count must be below 75,000
* Previously inserted Inferior Vena Cava Filter (IVC) filter.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All adults of at least 18 years of age who are to undergo sub-lobar resection, lobectomy, bilobectomy or pneumonectomy for lung cancer or metastatic lung disease will be offered the opportunity to participate in the study. The inclusion criteria are intentionally broad to increase the generalizability of the study. Eligibility criteria will be considered for enrollment in the study and are listed in the methodology section. The study population for both phases one and two of the study will have the same inclusion and exclusion criteria but will not include the same participants.
Sampling Method: Non-Probability Sample
Enrollment: 150 (Actual)
Dates: Start 2014-01; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
To determine the incidence of PE/DVT after lung resection for malignancies | 30 days post hospital discharge

SECONDARY OUTCOMES:
Incidence of post-operative PE and DVT comparing thoracotomy vs. VATS | 30 days post hospital discharge
Complications and mortality of DVT and PE post lung resection | 30 days post hospital discharge
Risk factors for the development of VTE post lung resection | 30 days post hospital discharge
Correlation between DVT and PE in patients developing PE | 30 days post hospital discharge
  In this specific population, many PE events might not be initiated by VTE, but rather by the result of in-situ arterial injury such as division, tying and/or clamping of the pulmonary artery branches during the lung resection. As a result, we postulate that we might identify patients with PE without a preceding DVT.

CONTACTS AND LOCATIONS:
Overall Officials: Yaron Shargall, MD BSc, Principal Investigator — St. Joseph's Healthcare Hamilton
Locations (2):
- Canada (2):
  - St. Joseph's Healthcare Hamilton, Hamilton, Ontario
  - Toronto General Hospital (UHN), Toronto, Ontario

REFERENCES:
- [Background] Geerts WH, Bergqvist D, Pineo GF, Heit JA, Samama CM, Lassen MR, Colwell CW. Prevention of venous thromboembolism: American College of Chest Physicians Evidence-Based Clinical Practice Guidelines (8th Edition). Chest. 2008 Jun;133(6 Suppl):381S-453S. doi: 10.1378/chest.08-0656. PMID 18574271
- [Background] Daddi G, Milillo G, Lupattelli L, Ragusa M, Lemmi A, Puma F, Agnelli G; Pulmonary Embolism in Thoracic Surgery Study Group. Postoperative pulmonary embolism detected with multislice computed tomography in lung surgery for cancer. J Thorac Cardiovasc Surg. 2006 Jul;132(1):197-8. doi: 10.1016/j.jtcvs.2006.03.036. No abstract available. PMID 16798341
- [Background] Kalweit G, Huwer H, Volkmer I, Petzold T, Gams E. Pulmonary embolism: a frequent cause of acute fatality after lung resection. Eur J Cardiothorac Surg. 1996;10(4):242-6; discussion 246-7. doi: 10.1016/s1010-7940(96)80146-1. PMID 8740059
- [Background] Dentali F, Malato A, Ageno W, Imperatori A, Cajozzo M, Rotolo N, Douketis J, Siragusa S, Crowther M. Incidence of venous thromboembolism in patients undergoing thoracotomy for lung cancer. J Thorac Cardiovasc Surg. 2008 Mar;135(3):705-6. doi: 10.1016/j.jtcvs.2007.10.036. No abstract available. PMID 18329505
- [Background] Ziomek S, Read RC, Tobler HG, Harrell JE Jr, Gocio JC, Fink LM, Ranval TJ, Ferris EJ, Harshfield DL, McFarland DR, et al. Thromboembolism in patients undergoing thoracotomy. Ann Thorac Surg. 1993 Aug;56(2):223-6; discussion 227. doi: 10.1016/0003-4975(93)91151-c. PMID 8347002
- [Background] Saarinen J, Kallio T, Sisto T, Tarkka M. Incidence of deep venous thrombosis after thoracotomy. Vasa. 2001 Nov;30(4):259-61. doi: 10.1024/0301-1526.30.4.259. PMID 11771209
- [Background] Cade JF, Clegg EA, Westlake GW. Prophylaxis of venous thrombosis after major thoracic surgery. Aust N Z J Surg. 1983 Aug;53(4):301-4. doi: 10.1111/j.1445-2197.1983.tb02451.x. PMID 6577843
- [Background] Azorin JF, Regnard JF, Dahan M, Pansart M. [Efficacy and tolerability of fraxiparine in the prevention of thromboembolic complications in oncologic thoracic surgery]. Ann Cardiol Angeiol (Paris). 1997 May-Jun;46(5-6):341-7. French. PMID 9295896
- [Background] Hull RD, Pineo GF, Stein PD, Mah AF, MacIsaac SM, Dahl OE, Butcher M, Brant RF, Ghali WA, Bergqvist D, Raskob GE. Extended out-of-hospital low-molecular-weight heparin prophylaxis against deep venous thrombosis in patients after elective hip arthroplasty: a systematic review. Ann Intern Med. 2001 Nov 20;135(10):858-69. doi: 10.7326/0003-4819-135-10-200111200-00006. PMID 11712876
- [Background] Bergqvist D, Benoni G, Bjorgell O, Fredin H, Hedlundh U, Nicolas S, Nilsson P, Nylander G. Low-molecular-weight heparin (enoxaparin) as prophylaxis against venous thromboembolism after total hip replacement. N Engl J Med. 1996 Sep 5;335(10):696-700. doi: 10.1056/NEJM199609053351002. PMID 8703168
- [Background] Planes A, Vochelle N, Darmon JY, Fagola M, Bellaud M, Huet Y. Risk of deep-venous thrombosis after hospital discharge in patients having undergone total hip replacement: double-blind randomised comparison of enoxaparin versus placebo. Lancet. 1996 Jul 27;348(9022):224-8. doi: 10.1016/s0140-6736(96)01453-5. PMID 8684199
- [Background] Comp PC, Spiro TE, Friedman RJ, Whitsett TL, Johnson GJ, Gardiner GA Jr, Landon GC, Jove M; Enoxaparin Clinical Trial Group. Prolonged enoxaparin therapy to prevent venous thromboembolism after primary hip or knee replacement. Enoxaparin Clinical Trial Group. J Bone Joint Surg Am. 2001 Mar;83(3):336-45. doi: 10.2106/00004623-200103000-00004. PMID 11263636
- [Background] Hull RD, Pineo GF, Francis C, Bergqvist D, Fellenius C, Soderberg K, Holmqvist A, Mant M, Dear R, Baylis B, Mah A, Brant R. Low-molecular-weight heparin prophylaxis using dalteparin extended out-of-hospital vs in-hospital warfarin/out-of-hospital placebo in hip arthroplasty patients: a double-blind, randomized comparison. North American Fragmin Trial Investigators. Arch Intern Med. 2000 Jul 24;160(14):2208-15. doi: 10.1001/archinte.160.14.2208. PMID 10904465
- [Background] Lassen MR, Borris LC, Anderson BS, Jensen HP, Skejo Bro HP, Andersen G, Petersen AO, Siem P, Horlyck E, Jensen BV, Thomsen PB, Hansen BR, Erin-Madsen J, Moller JC, Rotwitt L, Christensen F, Nielsen JB, Jorgensen PS, Paaske B, Torholm C, Hvidt P, Jensen NK, Nielsen AB, Appelquist E, Tjalve E, et al. Efficacy and safety of prolonged thromboprophylaxis with a low molecular weight heparin (dalteparin) after total hip arthroplasty--the Danish Prolonged Prophylaxis (DaPP) Study. Thromb Res. 1998 Mar 15;89(6):281-7. doi: 10.1016/s0049-3848(98)00018-8. PMID 9669750
- [Background] White RH, Romano PS, Zhou H, Rodrigo J, Bargar W. Incidence and time course of thromboembolic outcomes following total hip or knee arthroplasty. Arch Intern Med. 1998 Jul 27;158(14):1525-31. doi: 10.1001/archinte.158.14.1525. PMID 9679793
- [Background] Prandoni P, Falanga A, Piccioli A. Cancer and venous thromboembolism. Lancet Oncol. 2005 Jun;6(6):401-10. doi: 10.1016/S1470-2045(05)70207-2. PMID 15925818
- [Background] White RH, Zhou H, Romano PS. Incidence of symptomatic venous thromboembolism after different elective or urgent surgical procedures. Thromb Haemost. 2003 Sep;90(3):446-55. doi: 10.1160/TH03-03-0152. PMID 12958614
- [Background] Agnelli G, Bolis G, Capussotti L, Scarpa RM, Tonelli F, Bonizzoni E, Moia M, Parazzini F, Rossi R, Sonaglia F, Valarani B, Bianchini C, Gussoni G. A clinical outcome-based prospective study on venous thromboembolism after cancer surgery: the @RISTOS project. Ann Surg. 2006 Jan;243(1):89-95. doi: 10.1097/01.sla.0000193959.44677.48. PMID 16371741
- [Background] Bottaro FJ, Elizondo MC, Doti C, Bruetman JE, Perez Moreno PD, Bullorsky EO, Ceresetto JM. Efficacy of extended thrombo-prophylaxis in major abdominal surgery: what does the evidence show? A meta-analysis. Thromb Haemost. 2008 Jun;99(6):1104-11. doi: 10.1160/TH07-12-0759. PMID 18521515
- [Background] Kakkar VV, Balibrea JL, Martinez-Gonzalez J, Prandoni P; CANBESURE Study Group. Extended prophylaxis with bemiparin for the prevention of venous thromboembolism after abdominal or pelvic surgery for cancer: the CANBESURE randomized study. J Thromb Haemost. 2010 Jun;8(6):1223-9. doi: 10.1111/j.1538-7836.2010.03892.x. Epub 2010 Apr 30. PMID 20456751
- [Background] Bates SM, Jaeschke R, Stevens SM, Goodacre S, Wells PS, Stevenson MD, Kearon C, Schunemann HJ, Crowther M, Pauker SG, Makdissi R, Guyatt GH. Diagnosis of DVT: Antithrombotic Therapy and Prevention of Thrombosis, 9th ed: American College of Chest Physicians Evidence-Based Clinical Practice Guidelines. Chest. 2012 Feb;141(2 Suppl):e351S-e418S. doi: 10.1378/chest.11-2299. PMID 22315267
- [Background] Hurwitz LM, Yoshizumi TT, Goodman PC, Nelson RC, Toncheva G, Nguyen GB, Lowry C, Anderson-Evans C. Radiation dose savings for adult pulmonary embolus 64-MDCT using bismuth breast shields, lower peak kilovoltage, and automatic tube current modulation. AJR Am J Roentgenol. 2009 Jan;192(1):244-53. doi: 10.2214/AJR.08.1066. PMID 19098206
- [Background] Sodickson A, Baeyens PF, Andriole KP, Prevedello LM, Nawfel RD, Hanson R, Khorasani R. Recurrent CT, cumulative radiation exposure, and associated radiation-induced cancer risks from CT of adults. Radiology. 2009 Apr;251(1):175-84. doi: 10.1148/radiol.2511081296. PMID 19332852
- [Background] Venous thromboembolism: reducing the risk of venous thromboembolism (deep vein thrombosis and pulmonary embolism) in inpatients undergoing surgery. National Institute for Health and Clinical Excellence (NICE). 2010